CLINICAL TRIAL: NCT06460207
Title: A 4-day Study of Neurofeedback Training of Cognitive Control in Healthy Adults
Brief Title: Neurofeedback Removal of Emotional Information From Mind
Acronym: remtrain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Jarrod Lewis-Peacock, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01MH129042_remtrain; R01MH129042 (NIH)
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Neurofeedback; Cognitive Training; Memory, Short-Term; Functional Magnetic Resonance Imaging (fMRI)
Keywords: Suppression; Maintenance; Cognitive Control; Working Memory

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the positive or negative valence condition. They will encounter stimuli from their assigned valence only during the fMRI task, but from both valences during the behavioral tests, so that the investigators can evaluate whether any learning generalizes across emotional valence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive stimuli neurofeedback (Experimental): Participants will encounter only positive stimuli during the fMRI task but will be tested on both positive and negative valence stimuli during the behavioral memory tests.
  Interventions: Other: fMRI neurofeedback
- Negative stimuli neurofeedback (Experimental): Participants will encounter only negative stimuli during the fMRI task but will be tested on both positive and negative valence stimuli during the behavioral memory tests.
  Interventions: Other: fMRI neurofeedback

INTERVENTIONS:
Other: fMRI neurofeedback — fMRI neurofeedback is a technique that allows individuals to observe real-time feedback of their brain activity as measured by fMRI scans. During a session, the participant lies inside an MRI scanner while their whole brain is scanned. This data is processed in real-time by a computer and then presented to the participant in the form of visual feedback. This feedback might be presented as a graph, a color-coded representation, or some other easily interpretable format. The participant is instructed to modulate their brain activity based on the feedback they receive. This can involve various mental strategies, such as focusing attention on specific thoughts, images, or sensations. Over repeated sessions, participants learn to consciously influence their brain activity based on the feedback they receive. Through trial and error, they discover which mental strategies are most effective for achieving their desired changes in brain activity.

SUMMARY:
This project will examine whether individuals can be trained, using real-time feedback about brain function during neuroimaging, to effectively remove thoughts from mind by providing them with a sense of what it feels like to successfully remove a thought.

DETAILED DESCRIPTION:
On the first day, an anatomical MRI scan will be followed by a 12-min resting state scan, a 30-min item localizer task in which participants view a set of 80 scene stimuli 3 times each, and a 10-min memory test outside the scanner. The brain data from the localizer will be used to identify baseline measures of item-specific brain activity patterns. On 3 subsequent days (within the next 2 weeks), participants will receive neurofeedback training. In each 1-hr session, an anatomical scan will be followed by 8 runs (5 min each) of 20 trials, half with each operation, randomly ordered, and a 10-min behavioral memory test. In the scanner, participants will perform a working memory task in which they encode a scene image and then are instructed to either maintain that image in mind for a few seconds or to suppress that image from mind. At the end of each trial, neurofeedback will be provided to the participant visually to denote their "level of engagement" in the instructed operation on that trial. The neurofeedback is derived from the MRI classifier fit for the instructed operation (maintain or suppress) from a working memory operation classifier that is pre-trained on prior data. Participants (N=40) will be randomly assigned to either the positive or negative valence condition. They will encounter stimuli from their assigned valence only during the neuroimaging task, but from both valences during the behavioral tests, so that the investigators can evaluate whether any learning generalizes across emotional valence.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Speak English fluently
* Minimum 8th grade education
* Good hearing
* Good vision or minimal correction with contacts or eyeglasses

Exclusion Criteria:

* History of significant illnesses (including cardiovascular disease, cancer, immunodeficiency disorders (including HIV infection)
* Diabetes
* Unstable endocrine disorders
* Neurological disorders
* Neuromuscular disorders
* Blood dyscrasias
* History of major psychiatric disorders (including schizophrenia, bipolar disorder, and dementia)
* Substance dependence
* History of head trauma with loss of consciousness
* Cerebrovascular accident
* Seizures
* Neurosurgical intervention
* Metal implants in the body (including pacemakers, neurostimulators, or other metal objects)
* Metal piercings that cannot be removed for the scan
* Women who are pregnant or who think they may be pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neurofeedback learning | Within 2 weeks after the first day of the experiment, 3 neurofeedback training sessions lasting about 1 hour will occur at least 24 hours apart. The outcome measure will be computed at the end of all 3 sessions.
  Visual fMRI neurofeedback (e.g., the diameter of a circle) will be provided to the participant at the end of each trial denoting the "level of engagement" in the instructed operation on that trial. The neurofeedback score is derived from the fMRI pattern classifier using regularized logistic regression for the instructed operation from a pre-trained working memory operation classifier. Scores range from 0 to 1, with higher scores indicating better fits to the target pattern of activity. The investigators will quantify neurofeedback learning by computing changes in feedback scores within each session and across the sessions.
Neural consequences of control | Within 2 weeks after the first day of the experiment, 3 neurofeedback training sessions lasting about 1 hour will occur at least 24 hours apart. The outcome measure will be computed across all trials in each run, and for each of the 3 sessions.
  Proactive interference for the encoding of trial N, separately following maintain trials and suppress trials, will be assessed using within-subject item-specific activity pattern matching between the localizer data and the main task data. Proactive interference would be reflected in a reduced correspondence (lower scores) between the localizer representation for an item and the representation of that item when it is encoded on trial N. Higher scores would reflect a release from proactive interference.
Behavioral consequences of control | This outcome measure will be collected at the end of the first day of the experiment and at the end of each of the 3 subsequent neurofeedback sessions occurring at least 24 hours apart within the next 2 weeks.
  After each session, participants will be evaluated with behavioral memory tests on both positive and negative information. Two pictures (of the same valence) are presented for memorization on each trial, an instruction is given to manipulate the memory of one of those images, then a probe image appears and participants are to respond, as quickly and accurately as then can, YES if that probe image was one of the images presented at the beginning of the trial (even if the participant was asked to suppress that image) or NO otherwise. Half the probes contain new images. The accuracies and response times for this memory test will be statistically analyzed. The investigators will compare differences in these measures across condition (maintain vs. suppress) and cue type (manipulated vs. non-manipulated item). For the 3 neurofeedback sessions, the investigators will also relate a participant's neurofeedback scores with their behavioral performance on this memory test.

SECONDARY OUTCOMES:
Training transfer across valence | Within 2 weeks after the first day of the experiment, 3 neurofeedback training sessions lasting about 1 hour will occur at least 24 hours apart. This outcome measure will be collected at the end of each of the 3 sessions.
  The investigators will evaluate whether neurofeedback training transfers across emotional valence. Half of the participants will be trained on positive images, and half will be trained on negative images. The behavioral memory test at the end of each session includes both positive and negative images, and the outcomes measures from this test (as described in Primary Outcome 3) will be compared between these two groups of participants. Data will be statistically evaluated for whether the emotional valence on which a participant is trained has an effect that is selective (showing greater changes in accuracy and/or response times for trials of that same valence) or non-selective (no differences in performance metrics for trials with positive or negative valence).

CONTACTS AND LOCATIONS:
Overall Officials: Jarrod Lewis-Peacock, Ph.D., Principal Investigator — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the National Institutes of Mental Health Data Archive for all data collected in this experiment.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication of this study.

REFERENCES:
- [Background] Kim H, Smolker HR, Smith LL, Banich MT, Lewis-Peacock JA. Changes to information in working memory depend on distinct removal operations. Nat Commun. 2020 Dec 7;11(1):6239. doi: 10.1038/s41467-020-20085-4. PMID 33288756
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Banich MT, Mackiewicz Seghete KL, Depue BE, Burgess GC. Multiple modes of clearing one's mind of current thoughts: overlapping and distinct neural systems. Neuropsychologia. 2015 Mar;69:105-17. doi: 10.1016/j.neuropsychologia.2015.01.039. Epub 2015 Jan 28. PMID 25637772
- [Background] Lewis-Peacock JA, Kessler Y, Oberauer K. The removal of information from working memory. Ann N Y Acad Sci. 2018 Jul;1424(1):33-44. doi: 10.1111/nyas.13714. Epub 2018 May 9. PMID 29741212
- [Background] Lewis-Peacock JA, Drysdale AT, Oberauer K, Postle BR. Neural evidence for a distinction between short-term memory and the focus of attention. J Cogn Neurosci. 2012 Jan;24(1):61-79. doi: 10.1162/jocn_a_00140. Epub 2011 Sep 29. PMID 21955164
- [Background] Wang TH, Placek K, Lewis-Peacock JA. More Is Less: Increased Processing of Unwanted Memories Facilitates Forgetting. J Neurosci. 2019 May 1;39(18):3551-3560. doi: 10.1523/JNEUROSCI.2033-18.2019. Epub 2019 Mar 11. PMID 30858162